CLINICAL TRIAL: NCT01102296
Title: Division of Infectious Diseases, Department of Internal Medicine, National Taiwan University Hospital
Brief Title: Effectiveness of Hepatitis A Virus Vaccination Among Homosexual Males at Risk for Hepatitis A Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200903063M
Record Dates: First submitted 2010-01-08; First posted 2010-04-13 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis
Keywords: hepatitis A vaccine; male homosexual; HIV infection; male homosexuals who are seronegative for hepatitis A virus
MeSH Terms: conditions — Hepatitis; Homosexuality, Male; HIV Infections | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- male homosexuals (Active Comparator): HIV-uninfected male homosexuals will be provided 2 doses of HAV vaccine, which will be administered at baseline and 6th month of follow-up.
  Interventions: Biological: Hepatitis A vaccine
- HIV-infected male homosexuals, group1 (Active Comparator): HIV-infected male homosexuals will be provided 3 doses of HAV vaccine, which will be administered at baseline, 1st, and 6th month of follow-up.
  Interventions: Biological: Hepatitis A vaccine
- HIV-infected male homosexuals, group 2 (Active Comparator): HIV-infected male homosexuals will be provided 2 doses of hepatitis A vaccine, which will be administered at baseline and 6th month of follow-up.
  Interventions: Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: Hepatitis A vaccine — 2 or 3 doses of hepatitis A vaccine to HIV-infected male homosexuals and 2 doses of hepatitis A vaccine to HIV-uninfected male homosexuals.
  Other Names: HAVRIX (1440 ELISA unit)per dose.; MSM

SUMMARY:
Male homosexuals are at risk for hepatitis A virus (HAV) infection, and HAV vaccination has been recommended to prevent HAV infection in male homosexuals. HIV infection may impair serological responses to HAV vaccination in HIV-infected patients. The investigators hypothesize that 3 doses of HAV vaccine will improve serological responses to HAV vaccine in HIV-infected patients.

DETAILED DESCRIPTION:
In this study, we aim to compare the serological responses to HAV vaccination between HIV-infected patients who receive 2 doses or 3 doses of HAV vaccine and HIV-uninfected persons who receive 2 doses of HAV vaccine. Persons who identify themselves as male homosexuals aged younger than 40 years and are seronegative for hepatitis A virus will be enrolled. HAV vaccination will be provided free-of-charge. HIV-uninfected persons will receive 2 doses of HAV vaccine that will be administered at baseline and 6 months after the first dose, while HIV-infected patients will be given 2 doses or 3 doses of HAV vaccine; for those who choose to receive 3 doses, a second dose will be given 1 month after the first dose. A longitudinal follow-up of serological responses will be conducted to assess the effectiveness of HAV vaccination; HAV IgG will be determined at 6 months after the first dose of HAV vaccination(before the administration of the second dose), 12 months and 18 months after the first dose of HAV vaccination .

ELIGIBILITY:
Inclusion Criteria:

* Age between 18~40-years-old
* Homosexuals

Exclusion Criteria:

* Presence of symptoms or signs suggestive of active infection
* Allergy to vaccination
* Failure to provide written informed consent
* Use of immunosuppressive or immunomodulating agents or chemotherapy

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 582 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the proportion of vaccinees who achieve anti-HAV antibody concentrations of 20 mIU/ml or greater at week 48 of vaccination | 48 weeks

SECONDARY OUTCOMES:
the concentrations of anti-HAV antibody at week 48 of vaccination | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, MD, Principal Investigator — Division of Infectious Disease, Department of Internal Medicine, National Taiwan University Hopsital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan